CLINICAL TRIAL: NCT02098603
Title: Health Protection & Promotion for Oregon Correctional Officers
Acronym: DOC HEALTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency); Oregon Healthy Workforce Center (Unknown)
Responsible Party: Principal Investigator, Kerry Kuehl, Professor of Medicine, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: e7925; U19OH010154 (NIH)
Record Dates: First submitted 2013-10-07; First posted 2014-03-28 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Physical Activity; Nutrition; Health Promotion; Stress, Psychological; Metabolic Syndrome
MeSH Terms: conditions — Motor Activity; Stress, Psychological; Metabolic Syndrome | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Testing Only (No Intervention)
- Testing & Intervention (Experimental)
  Interventions: Behavioral: Testing & Intervention

INTERVENTIONS:
Behavioral: Testing & Intervention — Intervention involves a scripted peer-taught interactive curriculum, which is delivered as twelve, 30 minute weekly sessions incorporated into a team's usual work time or overtime activities.
  Arms: Testing & Intervention

SUMMARY:
More than 530,000 individuals work as US Correctional Officers (COs) responsible for overseeing the approximately 1.6 million offenders who are incarcerated at any given time in the United States. Prison work is regarded as one of the most difficult occupations with CO's having one of the highest nonfatal injury rates of all U.S. occupations. The few studies done on CO's show high levels of stress, cardiovascular disease, high job burnout, increased sick leave rates and absenteeism, and decreased quality of life leading to premature illness/injury and high employer healthcare costs. Many of these conditions could be prevented by specific training activities and healthier lifestyles. The investigators wish to test a worksite-based, health promotion curriculum in COs with the overall hypothesis that the program will improve health and decrease injuries. The program proposed would be the first occupational intervention to improve the safety, and emotional and physical health of those who are charged with the complex task of prison work protecting the investigators communities. If successful, this proposal would result in an exportable, practical occupational safety and health program applicable for use by local, state, and federal correctional facilities.

DETAILED DESCRIPTION:
Investigators will enroll up to 100 Correctional Officers from four Oregon Department of Corrections facilities for a randomized controlled 1-year assessment of the intervention. Participants will be evaluated at baseline, 6, and 12 months.

Primary study aims are; 1) Implement a randomized controlled efficacy trial of the Team-centered health promotion intervention, and assess its behavioral and occupational outcomes among COs, 2) Perform a cost analysis to determine the potential economic impact of this CO worksite health promotion program on illness/injury rates and disability claims, and 3) Determine relationships among specific intervention components with changes to behavior and occupational outcomes and assess by mediation analysis.

The intervention involves a scripted peer-taught interactive curriculum, which is delivered as twelve, 30 minute weekly sessions incorporated into a team's usual work time activities. The curriculum is designed to build understanding, healthy decision making skills and engender the social support of teammates; its content and scope reflects the core lifestyles activities used with fire fighters and law enforcement, along with adaptations for the needs of Correctional Officers in domains of the team-building, family support and psychological health.

Participant assessments include established survey instruments, physiological measures and selected laboratory parameters of outcomes and potential mediating variables at the individual, interpersonal and organizational levels. Intervention delivery and fidelity will be assessed. Multilevel and latent growth modeling and mediation analyses will be used to assess outcomes and the relationships among variables. At proposal completion there will be an evidenced-based, exportable occupational safety and health program for COs. Its critical components will be defined, and its benefits clearly determined.

ELIGIBILITY:
Inclusion Criteria:

* security employee of a participating facility in the Oregon Department of Corrections

Exclusion Criteria:

* none

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in BMI at 6 and 12 months | Baseline, 6 months, 12 months
  calculation of direct measurement of height and weight
Change from baseline in Fruit and Vegetable Intake at 6 and 12 months | Baseline, 6 months, 12 months
  questionnaire, NCI fruit/vegetables (Thompson et al., 2002)
Change from baseline in Physical Activity at 6 and 12 months | Baseline, 6 months, 12 months
  questionnaire; Elliot et al., 2007
Change from baseline in Stress at 6 and 12 months | Baseline, 6 months, 12 months
  questionnaire; Netemeyer RG et al, 1996; Cohen et al., 1983; Stanton et al, 2001
Change from baseline in Sleep at 6 and 12 months | Baseline, 6 months, 12 months
  questionnaire; Sorenson et al., 2011; Buysee et al., 1989; Buxton et al.; Rajaratnam et al., 2011
Change from baseline in Alcohol Use at 6 and 12 months | Baseline, 6 months, 12 months
  questionnaire
Change from baseline in Tobacco Use at 6 and 12 months | Baseline, 6 months, 12 months
  questionnaire; study specific development

SECONDARY OUTCOMES:
Change from baseline in Blood Pressure at 6 and 12 months | Baseline, 6 months, 12 months
  direct measurement
Change from baseline in Percent Body Fat at 6 and 12 months | Baseline, 6 months, 12 months
  direct measurement via Bioelectric Impedance Analysis scale
Change from baseline in Lipids and Lipoproteins at 6 and 12 months | Baseline, 6 months, 12 months
  direct measurement via Cholestech LDX analyzer
Change from baseline in Glucose at 6 and 12 months | Baseline, 6 months, 12 months
  direct measurement via Cholestech LDX analyzer
Cost-Effective Analysis | 12 months
  analysis of departmental aggregate data of injury rates and workers compensation claims

CONTACTS AND LOCATIONS:
Overall Officials: Kerry S Kuehl, MD, DrPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States